CLINICAL TRIAL: NCT00000327
Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment I(2)
Brief Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment I(2) - 2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11160-2; R01DA011160 (NIH); R01-11160-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: drug dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders

INTERVENTIONS:
Drug: Heroin Dependence

SUMMARY:
The purpose of this study is to compare the clinical efficacy of daily vs. 3-day (MWF) buprenorphine/naloxone combination tablet administration and determine whether outcomes are improved when using a 3-day schedule in which all doses are ingested at the clinic vs. one in which take-home doses are given on intervening days.

DETAILED DESCRIPTION:
Mon/Wed/Fri dosing with the 8 mg buprenorphine/naloxone tablet is as safe and effective as daily dosing and is preferred by patients to daily dosing. Multiple doses of the combination tablet (e.g. 16mg, 24mg) are well tolerated by patients. A 3 day schedule with take-outs is as effective as a 3-day schedule in which all medication is ingested at the clinic

ELIGIBILITY:
Inclusion Criteria:

Individual must be currently dependent and meet FDA criteria for narcotic maintenance treatment. Co-morbid substance abuse or dependence disorders may also be present. Individuals must be healthy despite drug dependency.

Exclusion Criteria:

Individuals with evidence of an active Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Axis I psychiatric disorder (e.g., psychosis, manic-depressive illness, organic psychiatric disorders), significant medical illness (e.g. liver or cardiovascular disease) or pregnant female subjects are excluded from study participation.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1997-06; Primary Completion 1997-08 (Actual); Study Completion 1997-08 (Actual)

PRIMARY OUTCOMES:
Drug use
Retention
Compliance
Dosing schedule preferences
Analog rating scale for dosing schedule effects

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Amass, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] Amass, L., Kamien, J.H., and Mikulich, S.K. Efficacy of and preference for 3-day vs daily dosing with the buprenorphine-naloxone combination tablet. presented to the 1998 Meeting of the College on Problems of Drug Dependence. Scottsdate, AZ (6/13-18). Presenting at CPDD 1998